CLINICAL TRIAL: NCT04505280
Title: Greater Occipital Nerve and Cervical Region Injection in Patients With Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cem Bölük, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-KAEK-2
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; Greater Occipital Nerve Block; Lidocaine
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): %1 lidocaine injections to greater occipital nerve and cervical region once a week for 4 weeks
  Interventions: Drug: Lidocaine 1% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine 1% Injectable Solution — Greater occipital nerve and cervical region injections once a week for 4 weeks

SUMMARY:
The aim of this study is to investigate the efficacy of greater occipital nerve block and cervical injections with lidocaine

DETAILED DESCRIPTION:
After being informed about the study and potantiel risks, all patients giving informed consent will undergo randomization in 1:1 ratio to 1% lidocaine or 0.9% saline groups

ELIGIBILITY:
Inclusion Criteria:

* Classical Trigeminal Neuralgia

Exclusion Criteria:

* Secondary Trigeminal Neuralgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Efficacy on pain severity | 3 months
  Efficacy on pain scores. Visual Analogue Scale (VAS). VAS is a ten-point scale where zero refers to no pain and ten refers to maximal pain
Efficacy on pain frequency | 3 months
  Pain frequency per day

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar University of Health Sciences, Afyonkarahisar, Kartal/Soğanlık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No